CLINICAL TRIAL: NCT05361512
Title: Characteristics of the Tsui Test and Pressure Waveform to Confirm Epidural Catheter Placement in Parturients With BMI ≥50 kg/m2
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 22-03
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Labor Pain
Keywords: epidural catheter; epidural analgesia; cesarean section; Tsui test; epidural waveform
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients having an epidural placed for labour analgesia or anesthesia for cesarean delivery: Patients with BMI>=50 who are having an epidural placed may take part in this study.
  Interventions: Device: Tsui test; Device: epidural waveform analysis

INTERVENTIONS:
Device: Tsui test — The stimulator is set at frequency of 1Hz with 0.2 msec pulse width and the current output ranging from 0 to 20 mA. The current output will be carefully increased from zero until motor activity is detected up to a maximum of 20 mA.
  Other Names: epidural electrical stimulation test (EEST)
Device: epidural waveform analysis — A pressurized 500ml normal saline bag will be connected to a pressure transducer kit and the transducer will be connected to a portable monitor with the scale set at 0-40 mmHg or to optimum scale. The transducer will be levelled with the heart approximated at the patient's manubrio-sternal angle, with the patient in the sitting position. Sterile tubing will be connected to the epidural needle and attached to transducer. The tubing connection will be filled with saline to ensure proper reflection of the pressure transducer tracing. Test will be considered positive in case of pulsatile waveform is observed in synchrony with heart rate.

SUMMARY:
The prevalence of obesity has increased worldwide, and the anesthetic care of patients with obesity remains a challenge for providers despite advances. Obesity during pregnancy is a risk factor for hypertensive disorders, gestational diabetes, emergency cesarean section and higher prevalence of difficult airway. Neuraxial techniques should always be preferred in women with obesity, particularly in those with body mass index (BMI) ≥50 kg/m2, where complications can be magnified. It is estimated an overall epidural failure rate of 4.3% in patients with obesity and an epidural failure rate of 13.7% in those with BMI ≥50 kg/m2. Hence, a confirmatory test of epidural catheter placement should prove useful in this patient population. The epidural electrical stimulation test (EEST) and the epidural waveform analysis are tests described in the literature as confirmatory methods for accuracy of placement of the epidural catheter.

The Tsui test has been well studied in obstetric patients, including required threshold electric currents and muscle contraction patterns. However, these studies have been conducted in patients receiving lumbar epidural catheters. Furthermore, they have not specifically included women with obesity class 3, particularly those with BMI≥50 kg/m2. In a recent study conducted in our department, the investigators have observed that patients with BMI≥50 kg/m2 require placement of an epidural catheter at a low-thoracic or high lumbar interspace, to allow the provision of effective surgical anesthesia for cesarean delivery, which often requires a modified incision, either transverse supra-umbilical or infra-umbilical. There are only few studies with waveform confirmation in obstetric patients showing conflicting results and certainly no studies under the circumstances described above. Finally, the Tsui test and the epidural waveform analysis have never been compared in the obstetric population.

The investigators aim to describe the characteristics of the Tsui test and of the epidural waveform analysis in parturients with BMI≥50 kg/m2 receiving epidural catheter placement at T12-L1 for both labor analgesia or anesthesia for cesarean delivery

DETAILED DESCRIPTION:
The Tsui test has been well studied in obstetric patients, including required threshold electric currents and muscle contraction patterns. However, these studies have been conducted in patients receiving lumbar epidural catheters. Furthermore, they have not specifically included women with obesity class 3, particularly those with BMI≥50 kg/m2. In a recent study conducted in our department, the investigators have observed that patients with BMI≥50 kg/m2 require placement of an epidural catheter at a low-thoracic or high lumbar interspace, to allow the provision of effective surgical anesthesia for cesarean delivery, which often requires a modified incision, either transverse supra-umbilical or infra-umbilical. There are only few studies with waveform confirmation in obstetric patients showing conflicting results and certainly no studies under the circumstances described above. Finally, the Tsui test and the epidural waveform analysis have never been compared in the obstetric population.

ELIGIBILITY:
Inclusion Criteria:

- Parturients with BMI≥50 kg/m2 requesting epidural labor analgesia or undergoing elective cesarean delivery

Exclusion Criteria:

* contraindication to epidural anesthesia
* allergy or hypersensitivity to lidocaine, bupivacaine or fentanyl
* those with implanted electronic devices.

Ages: 18 Years to 55 Years | Sex: Female
Age Groups: Adult
Study Population: Parturients with BMI≥50 kg/m2 requesting epidural labor analgesia or undergoing elective cesarean delivery.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Tsui test motor response: questionnaire | 15 minutes
  Tsui test motor response will be recorded as either: left, right or bilateral. Any increase in current requirement after the test dose will be recorded.
epidural waveform test (catheter) - questionnaire | 15 minutes
  A positive epidural waveform test through the catheter, defined as the presence of a pulsatile waveform observed in synchrony with heart rate: yes or no.

SECONDARY OUTCOMES:
epidural waveform test (needle) - questionnaire | 15 minutes
  A positive epidural waveform test though the needle, defined as the presence of a pulsatile waveform observed in synchrony with heart rate: yes or no
Tsui test motor response (before test dose): questionnaire | 15 minutes
  Tsui test motor response will be recorded as either: left, right or bilateral.
Tsui test current threshold (baseline) | 15 minutes
  Minimal electrical current required to produce a muscular contraction (mA) at baseline.
Tsui test current threshold (after test dose) | 15 minutes
  Minimal electrical current required to produce a muscular contraction (mA) 5 minutes after the test dose.
Laterality of the Tsui test: questionnaire | 15 minutes
  Laterality of the Tsui test, recorded as: unilateral right or left, or bilateral
Location of muscle group response to Tsui test: questionnaire | 15 minutes
  Muscle group responding to the electrical stimulation: abdominal wall, thigh, lower leg, foot (left or right)
Need for catheter mobilization: questionnaire | 15 minutes
  The need for catheter mobilization, including replacement (at any time after it is placed) will be documented as yes or no. The reason will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No